CLINICAL TRIAL: NCT04635241
Title: INHALEd Unfractionated HEParin for the Treatment of Hospitalised Patients With COVID-19 Meta-trial
Brief Title: Inhaled Heparin for Hospitalised COVID-19 Patients
Acronym: INHALE-HEP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Australian National University (Other)
Collaborators: Helwan University (Other); Clinica San Camilo, Argentina (Other); Frederick Health (Other); Dr Cipto Mangunkusumo General Hospital (Other); Dr. Moewardi General Hospital, Surakarta, Indonesia (Other); University of Sao Paulo (Other); St James Connolly Memorial Hospital (Other); University College Hospital Galway (Other); Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Frank van Haren, Professor, Australian National University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INHALE-HEP meta-trial
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Heparin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled heparin (Experimental): Inhaled nebulised unfractionated heparin in addition to standard care Dose 25,000 IU every 6 hours for up to 21 days
  Interventions: Drug: Unfractionated heparin
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Drug: Unfractionated heparin — Inhaled nebulised 6 hourly
  Arms: Inhaled heparin

SUMMARY:
This meta-trial is a prospective collaborative individual participant data meta-analysis of randomised controlled trials and early phase studies. Individual studies will be conducted in multiple countries, including Australia, the UK, the USA, Ireland, Argentina, Brazil and Egypt.

Adult patients admitted to the hospital with confirmed SARS-CoV-2 infection, who do not require immediate mechanical ventilation, will be randomised to inhaled nebulised heparin or standard care for up to 21 days or until the patient has no respiratory symptoms. All studies will collect a minimum core dataset. The primary outcome for the meta-trial is the proportion of patients who receive invasive mechanical ventilation censored at day 28. Individual studies may have specific outcome measures in addition to the core set.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital with COVID-19
* No immediate requirement for mechanical ventilation (points 3-5 on the WHO ordinal scale)
* Age equal to or greater than 18
* Able to provide informed consent

Exclusion Criteria:

* Pregnant women
* Known allergy to Heparin
* Participant in another clinical trial that is not approved for joint enrollment.
* APTT> 120 seconds, not due to anticoagulant therapy.
* Platelet count <20 x 109 per L
* Lung bleeding.
* Uncontrolled bleeding
* Advanced neurological impairment
* Advanced oncological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
Intubation rate | Day 28
  Proportion of patients requiring invasive mechanical ventilation

SECONDARY OUTCOMES:
WHO ordinal scale COVID19 | Day 7
  Number of patients showing 1 or 2 point worsening on the ordinal scale
Oxygenation | Day 7
  Daily ratio of partial pressure of oxygen to FiO2 (PaO2/FiO2)

CONTACTS AND LOCATIONS:
Overall Officials: Frank MP van Haren, MD, PhD, Study Chair — Australian National University
Locations (5):
- San Camilo Clinic, Buenos Aires, Argentina
- 15th May hospital, Cairo, Egypt
- Indonesia (3):
  - RS Universitas Indonesia, Depok
  - RSUP Dr Cipto Mangunkusumo, Jakarta
  - RSUD Dr Moewardi, Surakarta

IPD SHARING:
Plan to Share IPD: Undecided
This meta-trial is a prospective collaborative individual participant data meta-analysis of randomised controlled trials and early phase studies.

REFERENCES:
- [Background] van Haren FMP, Page C, Laffey JG, Artigas A, Camprubi-Rimblas M, Nunes Q, Smith R, Shute J, Carroll M, Tree J, Carroll M, Singh D, Wilkinson T, Dixon B. Nebulised heparin as a treatment for COVID-19: scientific rationale and a call for randomised evidence. Crit Care. 2020 Jul 22;24(1):454. doi: 10.1186/s13054-020-03148-2. PMID 32698853
- [Derived] van Haren FMP, Valle SJ, Neto AS, Schultz MJ, Laffey JG, Artigas A, Dixon B, Vilaseca AB, Barbera RA, Ismail TI, Mahrous RS, Badr M, DeNucci G, Sverdloff C, Camprubi-Rimblas M, Cosgrave DW, McNicholas B, Cody C, Curley G, Smoot TL, Staas S, Sann K, Sas C, Belani A, Hillman C, Manggala SK, Aditianingsih D, Sugiarto A, Yulianti M, Herikurniawan H, Sinto R, Auerkari AN, Permana SA, Woodcock A, Carroll M, Wilkinson T, Singh D, Shute JK, Carroll M, Page C. Efficacy of inhaled nebulised unfractionated heparin to prevent intubation or death in hospitalised patients with COVID-19: an investigator-initiated international meta-trial of randomised clinical studies. EClinicalMedicine. 2025 Sep 27;88:103339. doi: 10.1016/j.eclinm.2025.103339. eCollection 2025 Oct. PMID 41181828
- [Derived] van Haren FMP, Richardson A, Yoon HJ, Artigas A, Laffey JG, Dixon B, Smith R, Vilaseca AB, Barbera RA, Ismail TI, Mahrous RS, Badr M, De Nucci G, Sverdloff C, van Loon LM, Camprubi-Rimblas M, Cosgrave DW, Smoot TL, Staas S, Sann K, Sas C, Belani A, Hillman C, Shute J, Carroll M, Wilkinson T, Carroll M, Singh D, Page C. INHALEd nebulised unfractionated HEParin for the treatment of hospitalised patients with COVID-19 (INHALE-HEP): Protocol and statistical analysis plan for an investigator-initiated international metatrial of randomised studies. Br J Clin Pharmacol. 2021 Aug;87(8):3075-3091. doi: 10.1111/bcp.14714. Epub 2021 Jan 19. PMID 33377218